CLINICAL TRIAL: NCT06151015
Title: Testing the Combined Effect of Dietary Nitrate and Caloric Restriction on Cognitive and Vascular Function in Older Adults Living with Overweight or Obesity: a 28-Day Pilot Randomised Trial
Brief Title: The Combined Effect of Dietary Nitrate and Caloric Restriction on Cognitive and Vascular Function.
Acronym: CRNitrateMRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moira Taylor (Other)
Collaborators: King Abdulaziz University (Other)
Responsible Party: Sponsor-Investigator, Moira Taylor, Associate Professor, University of Nottingham
Organization: University of Nottingham (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 323-0723
Record Dates: First submitted 2023-11-06; First posted 2023-11-30 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Healthy; Older Adults; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Pilot, randomised, parallel trial
Masking Description: Whilst participants will not be actively told which arm they have been allocated to, they are likely to be aware that their energy requirement has not been met if they have been allocated to the calorie restricted group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dietary nitrate plus caloric restriction (Experimental): Participants will drink beetroot juice with a calorie-restricted diet for 28 days.
  Interventions: Other: Nitrate-rich beetroot juice plus calorie-restricted diet
- Dietary nitrate alone (Active Comparator): Participants will drink beetroot juice with a weight-maintenance diet for 28 days.
  Interventions: Other: Nitrate-rich beetroot juice plus weight-maintenance diet

INTERVENTIONS:
Other: Nitrate-rich beetroot juice plus calorie-restricted diet — One daily bottle (70ml) of nitrate-rich beetroot juice with a calorie-restricted diet (1,000kcal deficit).
  Arms: Dietary nitrate plus caloric restriction
Other: Nitrate-rich beetroot juice plus weight-maintenance diet — One daily bottle (70ml) of nitrate-rich beetroot juice with a weight-maintenance diet (energy will be met).
  Arms: Dietary nitrate alone

SUMMARY:
This pilot study will compare the effect of combining dietary nitrate and caloric restriction versus dietary nitrate alone. The participant will be contacted, having responded to an advertisement on social media and posters, to attend the screening visit. They will be asked about their health status, suitability for MRI and availability. The investigators will use physical activity and eating attitude questionnaires. The investigators will also measure their height, weight, body mass index (BMI), and blood pressure (BP) and undertake blood tests. If they are eligible, they will be randomised to one of the two arms. The first group will consume nitrate-rich beetroot juice with a calorie-restricted diet for 28 days. The second group will drink the same juice with a weight-maintenance diet for the same period. The food and drinks will be provided. The outcome measures will be measured twice (at the baseline and end visits) to evaluate the change. The primary outcome is the cognitive function. The secondary outcomes are peripheral vascular health (BP and microvascular perfusion), cerebral vascular health (brain blood flow), anthropometry, body composition, and exhaled NO and nitrate concentrations. Also, the feasibility and accessibility of the study will be assessed.

DETAILED DESCRIPTION:
Twenty healthy males and females, aged 60-70 years, non-smokers, and living with overweight or obesity (BMI 25-40 kg/m2) will be recruited to a 28-day pilot, randomised, parallel trial to follow one of the interventions (dietary nitrate with calorie-restricted diet or dietary nitrate with weight-maintenance diet) if they are eligible. Their energy requirement will be calculated using the Mifflin-St Jeor Equation, and the participant will be instructed to follow a healthy diet ( pre-diet standardisation) for three days before the intervention to minimise the effect of the sudden change of their habitual diet (during which their energy requirement will be met). At the Baseline Visit (Day 0), they will be randomised to one of the two arms, and the outcome measurements will be taken. Cognitive function will be measured via a pen-and-paper test (TMT) and a cognitive battery of tests (COMPASS). Clinic and home resting blood pressure (BP) will be measured using an automated BP monitor. Microvascular perfusion will be measured by a Laser Doppler monitor. Cerebral blood flow will be measured using a brain MRI scan. Height, weight, BMI, skinfold thickness, and waist circumference will be measured via a wall-mounted stadiometer, calibrated scale, BMI equation, calipers, and a tape measure, respectively. Body composition will be measured by a bioelectrical impedance analysis (BIA). Exhaled NO will be measured using a fractional exhaled nitric oxide analyser (FeNO). Blood samples will be taken to measure plasma nitrate concentrations. Physical activity will be monitored through a wearable smartwatch with an integrated accelerometer. The participants will be provided with 14 bottles of nitrate-rich beetroot juice (70 ml, which provides 6.5mmol of nitrate/day) with their allocated diet to be consumed in the next 14 days, starting from the next day (Day 1), and the remaining 14 days' supply will be delivered on Day 13. There will be an energy deficit of 1,000 kcal/day if they are allocated to the caloric restriction group. Otherwise, the energy requirement will be met. After completing the 28-day intervention, the participant will attend the End Visit (Day 29), to repeat the same study measurements they have done in the Baseline Visit. An exit feedback questionnaire will be given to collect information on the acceptability and compliance with the measurement protocols and intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able to give written informed consent for their participation in the study.
* Healthy.
* Non-smoking adults.
* Male or female.
* Aged 60 to 75 years.
* BMI between 25 and 40 kg/m2.

Exclusion Criteria:

* Systolic BP > 180mmHg and/or diastolic BP >110mmHg at the Clinic Screening Visit.
* Contraindication for MRI.
* Does not have adequate understanding of verbal and written information in English, sufficient to complete an MRI safety screening and to give informed consent.
* Any existing or previous medical condition that may affect the study outcomes (i.e., diabetes, kidney dysfunction, malignant cancer, brain surgery, stroke).
* Any medical treatment that may affect the study outcomes (i.e., diuretics, anti-acids, organic nitrates, anti-pyschotics or neuro-stimulants).
* Evidence of an eating disorder as indicated by the Three-factor eating questionnaire (Eating Attitudes Tests-26).
* Blood donation within the last 3 months of the anticipated intervention beginnings.
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance.
* High-alcohol consumers (≥ 14 units/week for females, and ≥ 22 units/week for males).
* Vegetarianism (likely to have very high nitrate intake and food provided during the dietary intervention unsuitable).
* Weight change over 3.0kg in the last 2 months (important influence on vascular function).

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Cognitive function (TMT-B) | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in cognitive function from the baseline after 28 days intervention using a pen-and-paper cognitive test (TMT-B) compared to the comparator.

SECONDARY OUTCOMES:
Composite score of cognitive function | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in the composite score of cognitive function from the baseline after 28 days intervention using a computerised cognitive battery (COMPASS) compared to the comparator.
Cognitive function individual tasks (alphabetic working memory) | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in the cognitive function of individual task (alphabetic working memory) from the baseline after 28 days of intervention using a computerised cognitive battery (COMPASS) compared to the comparator.
Cognitive function individual task (serial subtraction) | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in the cognitive function of individual task (serial subtraction) from the baseline after 28 days of intervention using a computerised cognitive battery (COMPASS) compared to the comparator.
Cognitive function individual task (stroop) | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in the cognitive function of individual task (stroop) from the baseline after 28 days of intervention using a computerised cognitive battery (COMPASS) compared to the comparator.
Cognitive function individual task (peg and ball) | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in the cognitive function of individual task (peg and ball) from the baseline after 28 days of intervention using a computerised cognitive battery (COMPASS) compared to the comparator.
Cognitive function individual task (simple reaction time) | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in the cognitive function of individual task (simple reaction time) from the baseline after 28 days of intervention using a computerised cognitive battery (COMPASS) compared to the comparator.
Cognitive function (TMT-A) | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in cognitive function from the baseline after 28 days intervention using a pen-and-paper cognitive test (TMT-A) compared to the comparator.
Clinic blood pressure for systolic and diastolic pressure | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in clinic blood pressure (systolic and diastolic pressure) from the baseline after 28 days intervention using automated blood pressure device compared to the comparator.
Continuous home blood pressure for systolic and diastolic pressure | Every three days starting from Day 1 until Day 28 of the intervention.
  Changes in home blood pressure (systolic and diastolic pressure) from the first day of the intervention until last day using an automated blood pressure device compared to the comparator.
Microvascular perfusion | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in microvascular perfusion from the baseline after 28 days intervention using a Laser Doppler monitor compared to the comparator.
Cerebral blood flow | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in cerebral blood flow from the baseline after 28 days intervention using a brain MRI scan compared to the comparator.
Anthropometry (weight) | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in weight in kilograms from the baseline after 28 days intervention using a calibrated scale compared to the comparator.
Anthropometry (BMI) | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in BMI in kg/m^2 from the baseline after 28 days intervention using the BMI equation (weight and height will be combined to report BMI in kg/m^2) compared to the comparator.
Anthropometry (skinfold thickness) | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in skinfold thickness in millimetre from the baseline after 28 days intervention using a skinfold calipers, compared to the comparator.
Anthropometry (waist circumference) | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in waist circumference from the baseline after 28 days intervention using a tape measure compared to the comparator.
Body composition (fat mass) | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in body composition (fat mass in kg) from the baseline after 28 days intervention using a bioelectrical impedance analysis (BIA) compared to the comparator.
Body composition (fat-free mass) | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in body composition (fat-free mass in kg) from the baseline after 28 days intervention using a bioelectrical impedance analysis (BIA) compared to the comparator.
Exhaled nitric oxide | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in nitric oxide from the baseline after 28 days intervention using a fractional exhaled nitric oxide analyser (FeNO) compared to the comparator.
Nitrate concentrations | Baseline Visit (Day 0)-one day before intervention, and End Visit (Day 29)-one day after intervention.
  Change in plasma nitrate concentrations from the baseline after 28 days intervention using an Ozone-based chemiluminescence compared to the comparator.
Feasibility and accessibility | End Visit (Day 29).
  A paper exit feedback questionnaire will be administered at the end of the study to collect information on the acceptability and compliance with the measurement protocols and intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Moira A Taylor, PhD RD, Principal Investigator — University of Nottingham
Locations (1):
- The University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only anonymised individual personal data will be shared, upon specific request from other researchers, for example, in order to undertake a meta analysis.
Supporting Information: Study Protocol, SAP
Time Frame: When requested.
Access Criteria: On receipt of requests, data will be made accessible if agreed by the University of Nottingham.

REFERENCES:
- [Background] Alharbi M, Stephan BC, Shannon OM, Siervo M. Does dietary nitrate boost the effects of caloric restriction on brain health? Potential physiological mechanisms and implications for future research. Nutr Metab (Lond). 2023 Oct 25;20(1):45. doi: 10.1186/s12986-023-00766-9. PMID 37880786
- [Background] Alharbi M, Chiurazzi M, Nasti G, Muscariello E, Mastantuono T, Koechl C, Stephan BC, Shannon OM, Colantuoni A, Siervo M. Caloric Restriction (CR) Plus High-Nitrate Beetroot Juice Does Not Amplify CR-Induced Metabolic Adaptation and Improves Vascular and Cognitive Functions in Overweight Adults: A 14-Day Pilot Randomised Trial. Nutrients. 2023 Feb 10;15(4):890. doi: 10.3390/nu15040890. PMID 36839248
- [Background] Babateen AM, Shannon OM, O'Brien GM, Olgacer D, Koehl C, Fostier W, Mathers JC, Siervo M. Moderate doses of dietary nitrate elicit greater effects on blood pressure and endothelial function than a high dose: A 13-week pilot study. Nutr Metab Cardiovasc Dis. 2023 Jun;33(6):1263-1267. doi: 10.1016/j.numecd.2023.02.024. Epub 2023 Mar 2. PMID 36958967
- [Background] Shannon OM, Gregory S, Siervo M. Dietary nitrate, aging and brain health: the latest evidence. Curr Opin Clin Nutr Metab Care. 2022 Nov 1;25(6):393-400. doi: 10.1097/MCO.0000000000000866. Epub 2022 Aug 9. PMID 35943128
- [Background] Siervo M, Babateen A, Alharbi M, Stephan B, Shannon O. Dietary nitrate and brain health. Too much ado about nothing or a solution for dementia prevention? Br J Nutr. 2022 Sep 28;128(6):1130-1136. doi: 10.1017/S0007114522002434. PMID 36688430
- [Background] Babateen AM, Shannon OM, O'Brien GM, Okello E, Smith E, Olgacer D, Koehl C, Fostier W, Wightman E, Kennedy D, Mathers JC, Siervo M. Incremental Doses of Nitrate-Rich Beetroot Juice Do Not Modify Cognitive Function and Cerebral Blood Flow in Overweight and Obese Older Adults: A 13-Week Pilot Randomised Clinical Trial. Nutrients. 2022 Mar 2;14(5):1052. doi: 10.3390/nu14051052. PMID 35268027
- [Background] Siervo M, Arnold R, Wells JC, Tagliabue A, Colantuoni A, Albanese E, Brayne C, Stephan BC. Intentional weight loss in overweight and obese individuals and cognitive function: a systematic review and meta-analysis. Obes Rev. 2011 Nov;12(11):968-83. doi: 10.1111/j.1467-789X.2011.00903.x. Epub 2011 Jul 18. PMID 21762426